CLINICAL TRIAL: NCT00664469
Title: INdians Followed for INtensive Lipid Lowering Treatment and Its safetY: To Assess The Safety And Effectiveness Of Ezetimibe Co-Administered With Any Statin Compared To Doubling Of Current Statin Daily Dose In South Asian Canadians
Brief Title: INdians Followed for INtensive Lipid Lowering Treatment and Its safetY
Acronym: INFINITY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry); Schering-Plough (Industry)
Responsible Party: Dr Mina Madan/Cardiologist, Schulich Heart Centre, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008_006; MK0653-153
Record Dates: First submitted 2008-04-01; First posted 2008-04-23 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EZE+statin (Experimental): ezetimibe 10 mg per day is added to actual statin regimen for 6 weeks followed by another 6 weeks if at goal or statin dose can be doubled.
  Interventions: Drug: ezetimibe
- Stat2 (Active Comparator): patients on statins has their dose doubled for 6 weeks followed by another 6 weeks in which ezetimibe is added or the statin dose is doubled again.
  Interventions: Drug: Comparator: Simvastatin 20, 40 and 80 mg; Drug: Comparator: Atorvastatin; Drug: Comparator: Rosuvastatin

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 10 mg/day over a 6-week course of treatment.
  Arms: EZE+statin
Drug: Comparator: Simvastatin 20, 40 and 80 mg — Simvastatin 20, 40 and 80 mg; actual statin regimen for 6 weeks followed by another 6 weeks if at goal or statin dose can be doubled.
  Arms: Stat2
Drug: Comparator: Atorvastatin — Atorvastatin 20, 40 & 80 mg; actual statin regimen for 6 weeks followed by another 6 weeks if at goal or statin dose can be doubled.
  Arms: Stat2
Drug: Comparator: Rosuvastatin — Rosuvastatin 10, 20 & 40 mg; actual statin regimen for 6 weeks followed by another 6 weeks if at goal or statin dose can be doubled.
  Arms: Stat2

SUMMARY:
In South Asian Canadians with documented coronary artery disease or diabetes and hypercholesterolemia with LDL-C levels > 2.0 mmol/L after 4 weeks of monotherapy with any statin: To compare the percent (%) of patients who achieve an LDL-C concentration of 2.0mmol/L after a 6-week course of treatment with ezetimibe 10 mg/day co-administered with any statin at any dose versus doubling of the current statin dose.

ELIGIBILITY:
Inclusion Criteria:

* According To The Judgment Of The Treating Physician, Changing Of The Current Regimen Or Doubling Of The Current Statin Dose Would Be Indicated For The Management Of The Patients Hypercholesterolemia
* All Women Of Childbearing Potential Must Be Practicing An Effective Method Of Contraception Beginning At Least Seven (7) Days Prior To The Study And Continuing At Least 14 Days After Study Completion Or After Study Discontinuation All Women Of Childbearing Potential Must Be Practicing An Effective Method Of Contraception Beginning At Least Seven (7) Days Prior To The Study And Continuing At Least 14 Days After Study Completion Or After Study Discontinuation
* Patient Is Male Or Female >= 18 Years Of Age
* Patient Is Of South Asian Descent, Specifically Canadian Citizens Or Landed Immigrants With Ethnic Background From India, Pakistan, Nepal, Bangladesh Or Sri Lanka.
* Patients With A Diagnosis Of Primary Hypercholesterolemia And Who Are Defined As Being "High Risk" With A Diagnosis Of Cad Or Diabetes, Either By Past Medical History Or By Angiographic Or Laboratory Evidence
* The Patient Has Serum Ldl-C > 2.0 Mmol/L While On Any Statin At Below Maximum (10 Mg, 20 Mg Or 40 Mg/Day) Daily Dose For A Minimum Of Four Weeks Prior To The Baseline Visit

Exclusion Criteria:

* Any Condition Which, In The Opinion Of The Investigator, Would Be Likely To Render The Patient Unable To Complete The Study Or For Which Study Participation Would Produce Significant Risk Or Not Be In The Best Interests Of The Patient
* Cancer Within The Past 5 Years (Except For Successfully Treated Basal And Squamous Cell Carcinoma)
* Disorders Of The Hematologic, Digestive (Including Malabsorptive Disorders), Or Central Nervous System Including Cerebrovascular Disease And Degenerative Diseases That Would Limit Study Evaluation Or Participation
* Doubling Of The Current Statin Dose Is Not Possible Due To Tolerability Or Safety Concerns Or Because The Patient Is Already On The Maximum Statin Dose (C.F. Individual Statin Monograph)
* Female Patient Receiving Hormone Therapy Not On A Stable Dose And Regimen For At Least 8 Weeks Prior To Visit 1 Or Is Unwilling To Continue The Same Regimen Throughout The Study
* History Of Mental Instability, Drug/Alcohol Abuse Within The Past 5 Years, Or Major Psychiatric Illness Not Adequately Controlled And Stable On Pharmacotherapy
* Individuals With Poor Mental Function, Drug Or Substance Abuse, Or Individuals With Unstable Psychiatric Illnesses, Which, In The Opinion Of The Investigator, May Interfere With Optimal Participation In The Study. Alcoholic Substance Abuse Would Be Defined As A Patient With Alcohol Consumption > 14 Drink Per Week. (A Drink Is: A Can Of Beer, Glass Of Wine, Or Single Measure Of Spirits)
* Medications That Are Potent Inhibitors Of Cyp3a4, Including Cyclosporin, Systemic Itraconazole Or Ketoconazole, Erythromycin, Telithromycin Or Clarithromycin, Nefazodone, Protease Inhibitors. In Addition, Patients Should Not Take Amiodarone, Verapamil, Or Danazol. Patient Is Consuming > 950ml (> 1 Quart) Of Grapefruit Juice/Day
* Non-Statin Lipid-Lowering Agents Including Fish Oils, Cholestin, Bile Acid Sequestrants, And Niacin (>200 Mg/Day) Taken Within 6 Weeks And Fibrates Within 8 Weeks Prior To Randomization At Visit 2 (Day 1)
* Oral Corticosteroids (Unless Used As Replacement Therapy For Pituitary/Adrenal Disease And On A Stable Regimen For At Least 6 Weeks Prior To Visit 1).
* Patient Has Liver Transaminases (Alt, Ast) > 50% Above The Upper Limit Of Normal At Screening (Visit 1) Or Active Liver Disease, And/Or Creatine Kinase (Ck) >50% Above The Upper Limit Of Normal (ULN)
* Patient Who Is Known Hiv Positive
* Patients Taking A Statin Medication Requiring Or Likely To Require Treatment With Prohibited Agents: Those With Known Interactions With Statins Including Antifungal Azoles (Itraconazole And Ketoconazole), Macrolide Antibiotics (Erythromycin And Clarithromycin), Nefazodone And Protease Inhibitors, Amiodarone And Verapamil
* Patients That Are Treatment Naive For Statins
* Patients Who Have Been Treated With Any Other Investigational Drug Within 30 Days Prior To Visit 1. (If < 30 Days, Contact The Clinical Monitor For A Case-By-Case Evaluation.)
* Serum Creatinine >2.0 Mg/Dl Or 177 Micromol/L At Screening Visit (Visit 1), Or Active Renal Disease With Significant Proteinuria (>1 Mg Albumin/Mg Creatinine), Or Nephrotic Syndrome At Visit 1
* Uncontrolled Endocrine Or Metabolic Disease Known To Influence Serum Lipids Or Lipoproteins (I.E. Secondary Causes Of Hyperlipidemia) Or Secondary Hypercholesterolemia Due To Hypothyroidism [T4 < 51.48nmol/L (< 4 Microg/Dl)] At Visit 1
* Use Of Therapeutic Doses Of Corticosteroids For Conditions Which, In The Opinion Of The Investigator, Are Likely To Require The Use Of Therapeutic Corticosteroid Therapy During The Subjects Period Of Participation In The Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary measure of efficacy will be the percentage of patients in each treatment arm achieving a target LDL-C > 2.0 mmol/L at week 6 assessment. This will be calculated as the percentage of patients achieving this end point at 6 weeks of treatment us | 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Merck Frosst Canada Ltd., Kirkland, Quebec, Canada